CLINICAL TRIAL: NCT03529812
Title: Exploring the Effect of Cognitively-Based Compassion Training (CBCT) on the Empathic Accuracy and Resilience of Spiritual Health Clinicians
Brief Title: CBCT for Spiritual Health Clinicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Jennifer Mascaro, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00098222
Record Dates: First submitted 2018-05-08; First posted 2018-05-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Health Behavior
Keywords: Behavioral intervention; Social intervention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: This study aims to enroll 30 hospital chaplain residents, 15 will have the CBCT intervention early and the other 15 will learn about CBCT later. Additionally, 500 patients who have spiritual services provided by the chaplains participating in the study will be enrolled in order to examine patient outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early-start group for CBCT-informed training (Experimental): Hospital chaplain residents receiving the Cognitively-Based Compassion Training (CBCT) education during the first unit of their year-long residency.
  Interventions: Behavioral: CBCT-informed training
- Delayed-start group for CBCT-informed training (Active Comparator): Hospital chaplain residents receiving the Cognitively-Based Compassion Training (CBCT) education midway through their year-long residency.
  Interventions: Behavioral: CBCT-informed training

INTERVENTIONS:
Behavioral: CBCT-informed training — Cognitively-Based Compassion Training (CBCT) is a secularized compassion meditation program adapted from the Tibetan Buddhist mind training (lojong) tradition. Lojong practices utilize a cognitive, analytic approach to challenge one's unexamined thoughts and emotions toward other people, with the long-term goal of developing altruistic emotions and behavior towards all people.

SUMMARY:
The Emory University Spiritual Health department will incorporate Cognitively-Based Compassion Training (CBCT) into their training curriculum beginning in Fall 2017, which provides the opportunity to compare students receiving the CBCT addendum with those receiving traditional chaplaincy training. This is a naturalistic study that examines the impact of incorporating CBCT into Emory's spiritual caregiver training program. The researchers will examine the effect of CBCT on empathic accuracy and resilience by comparing the first group of students who receive CBCT-informed training with chaplains who receive standard training in spiritual caregiving and receive CBCT later in the residency year. Comprehensive assessments will be conducted in order to examine whether outcomes for patients are improved for those receiving chaplain spiritual care augmented by CBCT compared to those receiving spiritual care from chaplains who receive CBCT later in their residency.

DETAILED DESCRIPTION:
Based on a wealth of research demonstrating the associations between physical health and psychosocial well-being, modern health care in the United States is characterized by an increasingly patient-centered model of care that places a premium on the holistic treatment of the patient as a physical, psychosocial, and spiritual whole. Hospital chaplains play a vital role in delivering emotional and spiritual care to a broad range of both religious and non-religious patients for a wide variety of stressors, and extensive research indicates that spiritual consults impact patient outcomes and satisfaction. However, there is remarkably little research on the "active ingredients" of chaplaincy spiritual care, and a subsequent lack of standardization and best-practice guidelines informing chaplain training and chaplain spiritual consulting. CBCT ® (Cognitively-Based Compassion Training) is a secularized compassion meditation program adapted from the Tibetan Buddhist mind training (lojong) tradition, and it may be an ideal addendum to both chaplain training programs and to the spiritual care consults provided by Emory University hospital chaplains to approximately 100,000 patients each year. This is a pilot study to explore the feasibility and impact of incorporating CBCT into the educational curriculum for chaplain residents. To this end, the researchers will (1) examine the impact of CBCT on burnout, compassion, and empathic accuracy among chaplains in training, (2) explore whether the impact persists through the end of the resident training, (3) evaluate the timing of the training within the existing curriculum to maximize its impact, (4) evaluate whether CBCT-informed interventions improve patient outcomes, and (5) explore chaplain and patient mediators of the impact of spiritual care consults on patient outcomes. Data acquired in this pilot study will be used to estimate efficacy and to inform a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria for Chaplains:

* Chaplain residents with Spiritual Health at Emory Healthcare

Inclusion Criteria for Chaplains:

* Patient of Emory Healthcare
* Requested a spiritual health consultation with a hospital chaplain

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Change in Depression Anxiety and Stress Scale (DASS) Score | Baseline, Week 5, Week 24, Week 29
  The Depression Anxiety and Stress Scale (DASS) is a 42-item likert-scale measure that assesses the frequency of symptoms of depression, anxiety and stress during the past week. Respondents indicate the degree to which they agree with each statement on a scale of 0 to 3 where 0 = does not apply to me at all and 3 = applied to me very much, or most of the time. Total scores range from 0 to 126 and higher scores indicate increased feelings of depression, anxiety and stress.
Change in Mental Health Continuum Short Form (MHC-SF) Score | Baseline, Week 5, Week 24, Week 29
  The Mental Health Continuum Short Form (MHC-SF) is a 14-item inventory assessing emotional well-being. Participants indicate how frequently they have experienced different feelings (such as feeling happy) in the past month. Responses are are a 6-point scale where 0 = never and 5 = every day. Total scores range from 0 to 70 and higher scores indicate greater well being.
Change in Professional Quality of Life Scale (ProQOL) Score | Baseline, Week 5, Week 24, Week 29
  The Professional Quality of Life Scale (ProQOL) is a 30-item inventory, the ProQOL is the most commonly used measure of the negative and positive effects of helping others who experience suffering. It has sub-scales for compassion satisfaction, burnout, and compassion fatigue. The sub-scales are summed and converted to t-scores with a mean of 50 and standard deviation of 10. Scores higher than 57 indicate professional satisfaction while scores below 40 indicate possible problems with feeling satisfied professionally.
Change in School-Burnout Inventory (SBI) Score | Baseline, Week 5, Week 24, Week 29
  The School-Burnout Inventory is a 9-item survey asking students about how much burnout, in the context of an academic environment, they have felt in the past month (for example, "I feel overwhelmed by my schoolwork"). Respondents indicate the degree to which they agree with each statement on a scale of 1 to 6 where 1 = completely disagree and 6 = completely agree. Total scores can range from 9 to 54, with higher scores indicating more burnout.
Change in Revised University of California, Los Angeles (UCLA) Loneliness Scale (R-UCLA) Score | Baseline, Week 5, Week 24, Week 29
  The Revised UCLA Loneliness Scale (R-UCLA) is a 20-item questionnaire measuring general feelings of social isolation and dissatisfaction with one's social interactions. Participants rate each item on a scale from 1 (never) to 4 (often). When scoring the scale, certain items are reversed so that low scores correspond with low loneliness. Total scores range from 20 to 80, where high scores indicate high feelings of loneliness.
Change in Empathic Accuracy (EA) Task Score | Baseline, Week 5, Week 24, Week 29
  The Empathic Accuracy (EA) Task is a dynamic video assessment that asks subjects to continuously rate the emotions of others as they tell emotional autobiographical stories. Empathic accuracy is the correlation between feelings of the story-tellers in the video and what the participants perceive the story-tellers feelings to be.
Change in Spiritual Meaning Scale (SMS) Score | Baseline, Week 5, Week 24, Week 29
  The Spiritual Meaning Scale (SMS) is a 15-item, likert-scale inventory that assesses the extent to which someone endorses a belief in something larger than themselves. Participants respond to statements like "life is inherently meaningful" on a scale of 1 to 5 where 1 = I totally disagree, 3 = I'm in between, and 5 = I totally agree. Certain items are scored in reverse. The total score ranges from 15 to 75 and higher scores indicate stronger belief.
Change in Jefferson Scale of Empathy Score | Baseline, Week 5, Week 24, Week 29
  The Jefferson Scale of Empathy is a 20-item scale designed to measure empathy in practicing health care professionals and health care professional students. Participants answer on a 7-point scale where 1 = strongly disagree and 7 = strongly agree. Total scores range from 20 to 140 where higher scores indicate increased empathy.

SECONDARY OUTCOMES:
National Comprehensive Cancer Network (NCCN) Distress Thermometer | Day 1 (before Spiritual Health consult)
  Patients will use the NCCN Distress Thermometer to rate levels of distress over the past week including the current day. The NCCN Distress Thermometer is a single-item screener of distress, with a scale from 0 (no distress) to 10 (extreme distress) represented through a visual graphic of a thermometer. Patients will complete the screening prior to having a Spiritual Health consult with the chaplain.
Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Emotions | Day 1 (after Spiritual Health consult)
  The PROMIS Self-Efficacy for Managing Emotions is a 15-item Likert scale self-report measure ("not at all confident"; "a little confident"; "somewhat confident"; "quite confident" and "very confident") completed by patients, which asks them to reflect on their own confidence levels in managing and controlling symptoms of anxiety, depression, helplessness, discouragement, frustration, disappointment, and anger. Raw scores range from 15 to 75 with higher scores indicating increased self efficacy. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
PROMIS Positive Affect | Day 1 (after Spiritual Health consult)
  The PROMIS Positive Affect questionnaire is a 15-item Likert-scale self-report measure completed by patients, which assesses momentary positive or rewarding affective experiences such as feelings and moods associated with pleasure, joy, elation, contentment, pride, affection, happiness, engagement, and excitement. Raw scores range from 15 to 75 with higher scores indicating increased positive feelings. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
Hospital Anxiety and Depression Scale (HADS) | Day 1 (after Spiritual Health consult)
  The Hospital Anxiety and Depression Scale (HADS) is a 14-item self-report questionnaire used to screen for the presence of depression and anxiety in physically ill patients. It is divided into two subscales: Anxiety (HADS-A) and Depression (HADS-D). Patients rate each item on a 4-point scale from 0 (absence) to 3 (extreme presence), with five of the 14 items reverse coded. Total scores range from 0 to 42, with higher scores indicating greater levels of anxiety and depression. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
PROMIS Emotional Support | Day 1 (after Spiritual Health consult)
  The PROMIS Emotional Support is a 4-item Likert-scale that assesses perceived feelings of being cared for and valued as a person. Each of the 4 questions has five response options ranging in value from one to five, with total scores ranging from 4 to 20. Higher scores indicate increased feelings of being supported emotionally. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
PROMIS Informational Support | Day 1 (after Spiritual Health consult)
  The PROMIS Informational Support is a 4-item Likert-scale that assesses perceived availability of helpful information or advice. Each of the 4 questions has five response options ranging in value from one to five, with total scores ranging from 4 to 20. Higher scores indicate increased perception of available information. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
PROMIS Social Isolation | Day 1 (after Spiritual Health consult)
  The PROMIS Social Isolation is a 4-item Likert-scale that assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. Each of the 4 questions has five response options ranging in value from one to five, with total scores ranging from 4 to 20. Higher scores indicate increased social isolation. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.
Scottish Patient Reported Outcome Measure (PROM) | Day 1 (after Spiritual Health consult)
  The Scottish Patient Reported Outcome Measure (PROM) is an 18-item self-report Likert-scale that assesses how a hospitalized patient perceived the Spiritual Care visit both during and after the consult. It also assesses the patient's present state regarding their situation and whether they view themselves as a spiritual or religious person. Responses range in value from 1 (not at all) to 5 (all of the time). Total scores range from 18 to 90 with higher scores suggesting increased positive feelings about the spiritual care received. Patients will complete the questionnaire after having a Spiritual Health consult with the chaplain.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Mascaro, PhD, Principal Investigator — Emory University
Locations (7):
- United States (7):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Wesley Woods Center, Atlanta, Georgia
  - St. Joseph's Hospital, Atlanta, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia